CLINICAL TRIAL: NCT04344080
Title: Effect of CytoSorb Adsorber on Hemodynamic and Immunological Parameters in Critical Ill Patients With COVID-19
Acronym: CYTOCOV-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYTOCOV-19; U1111-1250-2078 (Registry Identifier: UTN); DRKS00021199 (Registry Identifier: DRKS)
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: critically ill; intensive care medicine; CytoSorb; hemoadsorption
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CytoSorb-Therapy (Active Comparator): Therapy of COVID-19 with need for extracorporeal circulation (continuous renal replacement therapy or extracorporeal membrane oxygenation) using standard of care in Addition with hemoadsorption using CytoSorb-Adsorber
  Interventions: Device: CytoSorb-Therapy
- Standard of care (No Intervention): Therapy of COVID-19 with need for extracorporeal circulation (continuous renal replacement therapy or extracorporeal membrane oxygenation) using standard of care

INTERVENTIONS:
Device: CytoSorb-Therapy — Additional use of Cytosorb-Adsorber in patients with COVID-19 and need for extracorporeal circulation (continuous renal replacement therapy or extracorporeal membrane oxygenation)
  Arms: CytoSorb-Therapy

SUMMARY:
This prospective randomized single Center study investigates to what extent the physical elimination of the inflammatory mediators using the CytoSorb adsorber reduces the morbidity of severely and critically ill patients with Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID-19 disease
* refractory shock with need for norepinephrine ≥ 0.2 μg/kg/min for MAP ≥ 65 mmHg
* IL6 ≥ 500 ng/l
* Indication for CRRT or ECMO

Exclusion Criteria:

* Liver cirrhosis Child Pugh C
* "do not resuscitate"-order
* expected survival due to comorbidities < 14 days
* pregnancy or breastfeeding
* participation in another interventional trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a significant stabilization of hemodynamics for at least 24 hours | 24 hours
  Percentage of patients with a significant stabilization of hemodynamics ("shock reversal"), defined as a significant reduction of the noradrenaline dose (≤ 0.05 µg/kg/min) while maintaining mean arterial pressure ≥ 65 mmHg for at least 24 hours compared to control group

SECONDARY OUTCOMES:
Change in organ dysfunction | 10 days
  Change in organ dysfunction based on "Sequential Organ Failure Assessment" (SOFA) Score The SOFA score is made of 6 variables, each representing an organ system. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure) The worst physiological variables were collected serially every 24 hours of a patient's ICU admission. The "worst" measurement was defined as the measure that correlated to the highest number of points. The SOFA score ranges from 0 to 24.
Lactate clearance | 10 days
  Improving lactate clearance by lowering serum lactate levels
Renal replacement therapy | 10 days
  Time with need for renal replacement therapy
Extracorporeal Membrane Oxygenation | 10 days
  Time with Need for Extracorporeal Membrane Oxygenation
ICU length of stay | 90 days
  ICU length of stay
Time on mechanical ventilation | 10 days
  Time on mechanical ventilation
Cumulative catecholamine dose | 10 days
  Cumulative catecholamine dose
Overall and ICU mortality | 90 days
  Overall and ICU mortality
Change of plasma Interleukin-6 (IL6) level | 10 days
  Change of plasma Interleukin-6 (IL6) level
Change of plasma Interleukin-10 (IL10) level | 10 days
  Change of plasma Interleukin-10 (IL10) level
Change of plasma Procalcitonin (PCT) level | 10 days
  Change of plasma Procalcitonin (PCT) level
Change of HLA-DR level | 10 days
  Change of HLA-DR (Human Leukocyte Antigen - DR isotype) level of monocytes
Change of TNF alpha level after ex-vivo stimulation | 10 days
  Change of TNF-alfa level (Tumor Necrosis Factor alpha) level after LPS (Lipopolysaccharides) stimulation as sign of monocytic immunocompetence

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — University Hospital Hamburg-Eppendorf, Department of Intensive Care Medicine
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Published trial on PubMed.gov — https://pubmed.ncbi.nlm.nih.gov/36075200/